CLINICAL TRIAL: NCT07102095
Title: A Phase 1, Open-label, Single-dose Study to Assess the Influence of Hepatic Impairment on the Pharmacokinetics of of Sevabertinib (BAY 2927088)
Brief Title: A Study Evaluating How Moderate Liver Impairment Affects the Absorption, Distribution, Metabolism, and Elimination of Sevabertinib After a Single Oral Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 22988
Expanded Access: NCT06761976 (Available)
Record Dates: First submitted 2025-07-18; First posted 2025-08-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hepatic Insufficiency; Liver Diseases; Pharmacokinetics; Drug Metabolism
MeSH Terms: conditions — Hepatic Insufficiency; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Moderate Hepatic Impairment (Experimental): Approximately 10 participants with moderate impaired hepatic function (Child-Pugh B) to achieve approximately 8 evaluable participants
  Interventions: Drug: Sevabertinib
- Arm B: Normal Hepatic Function (Experimental): Approximately 10 matched control participants for Arm A with normal hepatic function
  Interventions: Drug: Sevabertinib

INTERVENTIONS:
Drug: Sevabertinib — Single oral dose of 20 mg sevabertinib administered as 2 x 10 mg film-coated tablets

SUMMARY:
This is a research study to understand how liver impairment affects the way the body processes a new cancer medicine called sevabertinib (BAY 2927088).

Sevabertinib is an experimental drug being developed to treat certain types of cancers that have specific genetic changes called HER2 mutations. This includes lung cancer, tumors that have spread to other parts of the body (metastatic), and tumors that cannot be removed with surgery (unresectable). Before this medicine can be given to cancer patients with liver problems, researchers need to understand how liver disease might change the way the body handles the drug.

The study will include about 20 people divided into two groups: 10 people with moderate liver problems (called Child-Pugh B liver impairment) and 10 healthy people with normal liver function. The healthy volunteers will be matched to the liver patients by age, sex, and weight to make fair comparisons.

All participants will take a single 20 mg dose of sevabertinib by mouth and stay in the research clinic for 5 days. During this time, researchers will take blood samples at specific times to measure how much drug is in the blood and how long it stays in the body. They will also monitor participants closely for any side effects.

The main goal is to see if people with liver problems have different drug levels in their blood compared to healthy people. This information will help doctors determine if cancer patients with liver disease need different doses of sevabertinib to be safe and effective.

The study will also look at the safety and tolerability of sevabertinib in both groups. Participants will have follow-up visits to ensure their continued health and safety.

This research is important because many cancer patients also have liver problems, and understanding how liver disease affects this new cancer treatment will help ensure it can be used safely and effectively in all patients who might benefit from it.

ELIGIBILITY:
Inclusion Criteria for all Participants:

* Participant must be 18 to 79 years of age inclusive, at the time of signing the informed consent.
* Normal hepatic function or moderate hepatic impairment.
* Body weight of at least 50 kg and BMI of within the range 18 to 40 kg/m2 inclusive.
* Female, of non childbearing potential only. Females must not be pregnant or breastfeeding, and must be documented as of non-childbearing potential (WONCBP). A negative pregnancy test is required.
* Male study participants of reproductive potential must agree to use adequate contraception when sexually active from signing the Informed Consent Form (ICF) until at least 3 months after the last dose of study intervention, and refrain from sperm donation during study intervention and for 3 months after the last dose of study intervention.
* Signed ICF.

Inclusion Criteria for Hepatic Impairment Group (Arm A)

* Documented liver disease with findings consistent with cirrhosis confirmed by histopathology, laparoscopy, fibroscan, CT, MRI, or ultrasound, AND
* Hepatic impairment (Child-Pugh B), AND
* Stable liver disease (i.e., same Child-Pugh class for at least 2 months prior to screening).

Inclusion Criteria for Normal Hepatic Function (Arm B)

* Have normal hepatic function, AND
* Fulfil Arm A matching criteria (sex, age, and body weight).

Exclusion Criteria for all Participants:

* Any existing relevant uncontrolled diseases of vital organs (e.g., heart, GI, pulmonary, or renal diseases), central nervous system (e.g., seizures), or other organs (e.g., uncontrolled diabetes mellitus [other than those related to hepatic impairment for the hepatically-impaired participants]) within 4 weeks prior to study intervention administration, including medically relevant infections and acute GI conditions (vomiting, diarrhea, and/or constipation).
* Known clinically relevant GI tract disorders (e.g., stomach ulcers, duodenal ulcers, GI bleeding, acute gastritis) or inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* Malignancy diagnosed or treated within the past 5 years (hepatocellular carcinoma within the past 2 years). Note: This does not include adequately-treated basal cell carcinoma or localized squamous cell carcinoma of the skin.
* Participants with primary or secondary biliary cirrhosis, or with sclerosing cholangitis.
* Pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination, and effects of the study intervention will be affected.
* Renal impairment with an eGFR ≤40 mL/min according to the CKD-EPI equation.
* Use of strong or moderate CYP3A4 inducers or inhibitors within 4 weeks or 5 half-lives prior to study intervention administration (whichever is longer) until last day of blood sampling for PK after study intervention administration.
* Use of drugs which may affect absorption, unless the drug is part of the mandatory dosing regimen for treatment of hepatic impairment or related conditions.
* Use of supplements or herbal remedies within 2 weeks prior to the first study intervention administration (except for vitamin supplementation).
* Use of anti-coagulant drugs.
* Positive alcohol blood/urine test at screening.
* Positive blood/urine drug screening indicating drug abuse (except for participants with hepatic insufficiency on an approved prescription for opioids or benzodiazepines who agree to withhold the use of opioids or benzodiazepines from 12 hours pre- and 12 hours post-intervention administration).
* Insufficiently controlled diabetes mellitus with HbA1c >10% within 6 months prior to study intervention administration.
* Consumption of food and beverages containing grapefruit, Seville orange, tangelo, or pomelos within 2 weeks prior to study intervention administration and up to the last PK sampling.
* Special diets preventing the participants from eating the standard meals during the study or unwillingness to eat the standard meals during the study.
* Use of recreational drugs, with the exception of cannabis (see below), carnitine products, anabolics, or high dose vitamins (except for medication against vitamin deficiency in hepatic impairment).

Cannabis containing products should be stopped 5 days prior to study intervention and should not be used during the in-house period of the study until after participant discharge from the clinic.

- Smoking more than 10 cigarettes daily (including vaping equivalent to approximately 10 cigarettes daily), or, unwilling to refrain from smoking and/or vaping from 22:00 on the day prior to study intervention administration and on Day 1 until 12 hours after study intervention administration.

Exclusion Criteria for Hepatic Impairment Group (Arm A) Medical Conditions

* Ascites qualitatively estimated as severe or requiring acute or frequent paracentesis (no emptying and/or albumin supplementation required within 30 days prior to Day 1 [or at least within 14 days], or during the course of the study, as judged by the investigator), or a recent history of paracentesis.
* Encephalopathy of Grade >2. Examinations
* ALP ≥4 × ULN.
* AST, ALT or GGT ≥4 × ULN.
* Platelet count <60 × 10^9/L.
* Hemoglobin <9 g/dL.
* Serum albumin <2 g/dL.
* INR >2.3.

Exclusion Criteria for Normal Hepatic Function (Arm B)

* Increase of liver enzymes (e.g., ALT, AST, GGT, or total bilirubin) above ULN.
* Increase of lipase and amylase (except isolated marginal increases of lipase or amylase to account for variability of the parameters, and the participant is asymptomatic and has no other laboratory changes assuming disease based on medical judgment).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2025-07-24 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve (AUC) of sevabertinib | 0-96 hours post-dose
  To assess the influence of hepatic impairment on sevabertinib exposure. AUC from time zero to the last data point larger than the lower limit of quantification (LLOQ) (AUC(0-tlast) and the unbound AUC(0-tlast) will be used as the main parameters if AUC cannot be reliably determined in all participants.
Unbound area under plasma concentration-time curve AUC (AUCu) of sevabertinib | 0-96 hours post-dose
  To assess the influence of hepatic impairment on sevabertinib exposure. AUC from time zero to the last data point larger than the lower limit of quantification (LLOQ) (AUC(0-tlast) and the unbound AUC(0-tlast) will be used as the main parameters if AUC cannot be reliably determined in all participants.
Maximum observed drug concentration (Cmax) of sevabertinib in plasma | 0-96 hours post-dose
  To assess the influence of hepatic impairment on sevabertinib exposure.
Unbound Cmax (Cmax,u) of sevabertinib in plasma | 0-96 hours post-dose
  To assess the influence of hepatic impairment on sevabertinib exposure.

SECONDARY OUTCOMES:
Incidence and severity of adverse events | From signing of informed consent form (ICF) until follow-up visit (approximately 2 weeks).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami - Oncology, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No
Currently, there is no established plan for the sharing of Individual Patient Data (IPD) from this study. The availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA 'Principles for responsible clinical trial data sharing.' This pertains to the scope, timepoint, and process of data access.
  As such, Bayer commits to considering requests from qualified researchers for patient- / study-level clinical trial data, and documents from clinical trials involving medicines and indications approved in the US and EU. However, this commitment does not reflect an active IPD sharing plan. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Researchers can use www.vivli.org to request access to IPD and documents from clinical studies to conduct research. Information on Bayer's criteria for listing studies is provided in the member section of the portal.